CLINICAL TRIAL: NCT06128005
Title: Evaluate Knowledge Translation Care Plan on Knowledge, Attitude, and Practice of Caregivers and Care Effects of Patients With Pressure Injury
Brief Title: Pressure Injury、Caregiver、Knowledge Translation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yi-Syuan Lai (Other)
Responsible Party: Sponsor-Investigator, Yi-Syuan Lai, nurse, National Defense Medical Center, Taiwan
Organization: National Defense Medical Center, Taiwan (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: pressureinjury853121
Record Dates: First submitted 2022-04-11; First posted 2023-11-13 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Pressure Injury; Pressure Ulcer
Keywords: caregiver; nursing plan
MeSH Terms: conditions — Pressure Ulcer | interventions — Nursing

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- knowledge translation in nursing for pressure injury care (Experimental): Using guideline and evidence based practice for pressure injury. The experimental group has received knowledge translation in nursing for pressure injury care with precaution teaching plan by using self-designed teaching materials, manuals, videoes, multimedia tools (power point, LINE official account, LINE one-on-one lesson, virtual lesson), in-person assistance and assessment in 12weeks.
  Interventions: Behavioral: knowledge translation in nursing for pressure injury care
- Regular care (Placebo Comparator): The controlled group maintained the regular nursing intervention.
  Interventions: Behavioral: knowledge translation in nursing for pressure injury care

INTERVENTIONS:
Behavioral: knowledge translation in nursing for pressure injury care — Pressure injury's knowledge and healing of wound.

SUMMARY:
Background and importance:

In 2003, a pressure injury is listed as one of the indicators of care quality in clinical setting by Taiwan joint commission on hospital accreditation. That reflects that a pressure injury is a significant heath care issue. Nowadays, it still constantly happens at hospitals, home, and nursing homes: Pressure injuries cause pain, and increase length of hospital stay, rehospitalization rate, and death rate. In current clinical practice, standardized guidelines and basic principles are followed for pressure injury management, and it is found that most of the caregivers are unsure about what are the consequences of having pressure injuries and how to manage and prevent them. Therefore, the caregivers are more passive, and feel nervous and confused. In literature, there are guidelines for pressure injury prevention and management. However, they are primarily designed for heath professionals. As a result, to achieve evidence-based practice and knowledge translation, I hope to make individual management plans for each patient, provide caring support, and follow up with patients. And caregivers can benefit from knowledge, attitude, practice, and caring effect.

DETAILED DESCRIPTION:
Goals:

The study aims to achieve knowledge translation in nursing for pressure injury care. The caregivers of patients with pressure injuries and their family can benefit from translating of knowledge, attitude, and practice, and they can have more knowledge related to pressure injuries, and learn how to react to and care for patients. In this way, it will be possible to promote wound healing and prevent recurrence of pressure injuries.

Method:

This study is a randomized controlled trial. There are seventy participants. The experimental group receives care plans in which knowledge translation is applied, and the control group receives usual care. Generalized estimating equations, GEE, is used to assess the effectiveness of care plans with knowledge translation for patients and family with pressure injuries.

ELIGIBILITY:
Inclusion Criteria:

1. Grade 1-3 pressure injury diagnosed by medical staff.
2. The patient needs to have a caregiver.
3. The patient and the caregiver need to be older than 20 years old, (4) The informed consent of this study.

(5) The caregiver Those who understand the content of health education (MMSE>24 points)

Exclusion Criteria:

1. The patient has >3 disease diagnoses,
2. The patient is diagnosed by a doctor as a terminally ill patient or the life expectancy is less than 3 months,
3. There is a life-threatening acute problem (active bleeding site, acute myocardial infarction, acute bronchitis, etc. ),
4. pressure injury caused by invasive pipeline placement,
5. need to wear non-invasive positive pressure respirator, (6) need to stay in intensive care center for a long time (>10 days),
6. need a long time For surgical patients, each operation takes > 5 hours,
7. the caregiver has dementia,
8. the caregiver has mental illness or alcohol and drug addiction,
9. no caregiver.

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-03-02 (Actual); Study Completion 2024-06-02 (Estimated)

PRIMARY OUTCOMES:
wound healing | 6 weeks and 12 weeks
  PUSH tool. Measure Length x Width, Exudate Amount and Tissue Type in pressure injury.
caregiver's knowledge | 6 weeks and 12 weeks
  Using a self-made questionnaire, the informal caregivers' knowledge of pressure injuries, such as: how does a pressure injury form, what are the care methods for a pressure injury, what should be prepared for wound care, methods to prevent a pressure injury, etc.
caregiver's attitude | 6 weeks and 12 weeks
  Use the self-made questionnaire to understand the caregivers' attitudes towards pressure injuries, such as whether they have motivation to care for them, whether they think it is important to prevent pressure injuries, whether they are confident that they can take good care of them, etc.
caregiver's practice | 6 weeks and 12 weeks
  Using a self-made questionnaire, the caregiver actually evaluates the situation of caring for the crush injury, such as: body positioning, repositioning, nutritional supply status, wound dressing change, wound grading assessment, body cleanliness, whether the protrusion of the bone is paid attention to, reducing Pressure equipment, etc.

SECONDARY OUTCOMES:
The recurrence rate of pressure injury three months after intervention | 12 weeks
  Patients with reoccurrence of pressure injury/Total number of experimental group or control group*100%
The rehospitalization rate | 12 weeks
  Number of patients re-admitted for pressure injuries /Total number of experimental group or control group *100%
The mortality rate | 12 weeks
  The number of Patient deaths/Total number of experimental group or control group *100%

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Syuan Lai, Study Chair — Student
Locations (1):
- Vivian, Keelung, Zhongzheng District, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Evaluate on the wound healing, knowledge and caring behaviors of hospitalized patients with pressure injury
Supporting Information: CSR
Time Frame: When I will complete the research, that can be sharing forever.
Access Criteria: Anyone have pressure injury's problem

REFERENCES:
- [Background] Santamaria N, Gerdtz M, Sage S, McCann J, Freeman A, Vassiliou T, De Vincentis S, Ng AW, Manias E, Liu W, Knott J. A randomised controlled trial of the effectiveness of soft silicone multi-layered foam dressings in the prevention of sacral and heel pressure ulcers in trauma and critically ill patients: the border trial. Int Wound J. 2015 Jun;12(3):302-8. doi: 10.1111/iwj.12101. Epub 2013 May 27. PMID 23711244
- [Background] Munoz N, Posthauer ME, Cereda E, Schols JMGA, Haesler E. The Role of Nutrition for Pressure Injury Prevention and Healing: The 2019 International Clinical Practice Guideline Recommendations. Adv Skin Wound Care. 2020 Mar;33(3):123-136. doi: 10.1097/01.ASW.0000653144.90739.ad. PMID 32058438
- [Background] Mervis JS, Phillips TJ. Pressure ulcers: Pathophysiology, epidemiology, risk factors, and presentation. J Am Acad Dermatol. 2019 Oct;81(4):881-890. doi: 10.1016/j.jaad.2018.12.069. Epub 2019 Jan 18. PMID 30664905
- [Background] Lin F, Wu Z, Song B, Coyer F, Chaboyer W. The effectiveness of multicomponent pressure injury prevention programs in adult intensive care patients: A systematic review. Int J Nurs Stud. 2020 Feb;102:103483. doi: 10.1016/j.ijnurstu.2019.103483. Epub 2019 Nov 21. PMID 31835122
- [Background] Jeyathevan G, Cameron JI, Craven BC, Jaglal SB. Identifying Required Skills to Enhance Family Caregiver Competency in Caring for Individuals With Spinal Cord Injury Living in the Community. Top Spinal Cord Inj Rehabil. 2019 Fall;25(4):290-302. doi: 10.1310/sci2504-290. PMID 31844381
- [Background] Tescher A, Deppisch M, Munro C, Jorgensen V, Cuddigan J. Perioperative pressure injury prevention: National Pressure Injury Advisory Panel root cause analysis toolkit 3.0. J Wound Care. 2022 Dec 1;31(Sup12):S4-S9. doi: 10.12968/jowc.2022.31.Sup12.S4. PMID 36475846
- [Background] Haesler E, Pittman J, Cuddigan J, Law S, Chang YY, Balzer K, Berlowitz D, Carville K, Kottner J, Litchford M, Moore Z, Mitchell P, Sigaudo-Roussel D. An exploration of the perspectives of individuals and their caregivers on pressure ulcer/injury prevention and management to inform the development of a clinical guideline. J Tissue Viability. 2022 Feb;31(1):1-10. doi: 10.1016/j.jtv.2021.10.008. Epub 2021 Oct 30. PMID 34776327
- [Background] Cuddigan J, Haesler E, Moore Z, Carville K, Kottner J. Development, dissemination and evaluation of a smartphone-based app for pressure ulcer/injury prevention and treatment for use at the bedside. J Wound Care. 2022 Dec 1;31(Sup12):S29-S39. doi: 10.12968/jowc.2022.31.Sup12.S29. PMID 36475841